CLINICAL TRIAL: NCT05394883
Title: The SPROUT (Pilot) Project: Starting Pregnancy With Robustness for Optimal Upward Trajectories
Brief Title: The SPROUT (Pilot) Project
Acronym: SPROUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Erin Wentz PT PhD PCS, Assistant Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPROUT
Record Dates: First submitted 2022-05-03; First posted 2022-05-27 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy Related; Infant Development; Adherence, Treatment; Activity, Motor
Keywords: pregnancy; supervised exercise; home exercise; fitness; maternal health outcomes; neonatal outcomes; feasibility; adherence
MeSH Terms: conditions — Treatment Adherence and Compliance; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a pilot investigation (feasibility) of a future larger study of interventional design with randomization. Participants in the pilot phase of the project will be randomized into one of three groups: supervised exercise, home exercise, or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Exercise (Experimental): Women randomized to Supervised Exercise group will attend two to three exercise classes/week.
  Interventions: Behavioral: Supervised Exercise
- Home Exercise (Experimental): Women assigned to Home Exercise group will receive instructions for their home walking and exercise program.
  Interventions: Behavioral: Home Exercise
- Usual Care (No Intervention): The Usual Care group will receive an exercise log to record any weekly activity in addition to a weekly phone call/text/email to remind the individual to complete the weekly exercise log.

INTERVENTIONS:
Behavioral: Supervised Exercise — Women randomized to Supervised Exercise group will attend two to three exercise classes/week. Each session will consist of: 5-min flexibility warm-up and cool-down; 40 min of moderate intensity calculated as 40-59% Heart Rate Reserve (HRR) along with Rating of Perceived Exertion (RPE) between 13-14; and 20 minutes of resistance with an additional 30 minutes of unsupervised home aerobic activity per week. The women will be given their choice of aerobic equipment or walking either track/ treadmill to achieve a total of 40 minutes of moderate intensity exercise. The Supervised Exercise group will receive exercise counseling during their first meeting in addition to materials on the benefits of exercise, a log to record additional activity completed each week, goal setting, making time for exercise/making exercise a habit and exercise behavioral strategies.
  Arms: Supervised Exercise
Behavioral: Home Exercise — Women assigned to Home Exercise group will receive instructions for their home walking program including tips for walking indoors and outdoors, exercise handouts for warm-up/cool-down activities, demonstrations for resistance training activities and an exercise log. Women assigned to Home Exercise group will be contacted once per week to discuss their progress, barriers/challenges faced, ask questions, and strategies to achieve the exercise guidelines. The Home Exercise group will receive exercise counseling during their first meeting in addition to materials on the benefits of exercise, a log to record additional activity completed each week, goal setting, making time for exercise/making exercise a habit and exercise behavioral strategies.
  Arms: Home Exercise

SUMMARY:
The purpose of this research is to study two different approaches to exercise during pregnancy that investigators believe will result in improved health for moms and babies. The investigators are trying to determine if the two types of exercise programs (supervised & home exercise) result in health improvements for moms and babies. The investigators also want to see if the tests and questionnaires used in the study can detect changes in a mom's aerobic fitness, quality of life (QOL), fatigue, sleep quality, depression, and weight change throughout pregnancy and 6-months after birth.

DETAILED DESCRIPTION:
Historically, pregnant women were advised to refrain from exercise due to concerns of maternal and fetal risk such as preterm delivery, low infant birth rate and fetal stress. Despite current research that has demonstrated substantial benefits for maternal, fetal, and infant health, only 9-15% of pregnant women meet the current physical activity recommendations. In addition, pregnancy exercise research is confounded by a lack of randomized controlled trials (RCT) that include diversity in participant demographics, specifically inner city populations, and difficulty accurately quantifying weekly exercise volume. The investigators propose a pilot RCT investigating two different approaches to exercise intervention across a spectrum of demographics that the investigators believe will result in improved exercise adherence as well as in maternal and infant health outcomes. Specific Aim #1: To determine the feasibility of two types of exercise interventions (supervised & home exercise) in terms of design, implementation and adherence. Our working hypothesis is that both supervised and home exercise interventions will be implementable as designed in pregnant women as evidenced by recruitment, eligibility, retention, follow-up and exercise adherence from 1st trimester through 6-months post-natal at a 60% rate, but that adherence to the two types of exercise interventions will differ by demographic. A secondary exploratory hypothesis is that the investigators will be able to successfully recruit and retain 50% of our pregnant women from the Syracuse Community Health Center (primarily women with lower resources). Specific Aim #2: To determine the appropriateness of the outcome measures proposed for the exercise intervention in detecting changes in maternal aerobic fitness, quality of life (QOL), fatigue, sleep quality, depression, and weight change throughout pregnancy and 6-months post-natal as measured by the Balke Ware submaximal test; SF-12 Generic Quality of Life (QOL); Multidimensional Fatigue Inventory (MFI); Pittsburgh Sleep Quality Index (PSQLI); Center for Epidemiologic Studies Depression Scale (CES-D); Edinburgh Postnatal Depression Scale (EPDS); and the Pregnancy Physical Activity Questionnaire (PPAQ). Our working hypothesis is that the above outcome measures will be able to detect changes in maternal outcome measures in both exercise groups. Because this is a feasibility study, the results will be used as preliminary data to apply for future funding and also will provide variable quantitative and qualitative data for validating interventions that can increase adherence to exercise guidelines during pregnancy in women with different ethnic and socioeconomic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women (i.e. 18 years of age and older)
* Low risk, singleton pregnancy
* In first trimester of pregnancy (6 to 13 weeks gestation)
* Without absolute contraindications to moderate intensity exercise during pregnancy as defined by the American College of Obstetricians and Gynecologists
* Exercise clearance from OB/GYN

Exclusion Criteria:

* Pregnancies greater than low risk for any reason
* Pregnant with more than one fetus
* Absolute exercise contraindications and/or lack of exercise clearance from OB/GYN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
The Bayley Scales of Infant Development, 4th edition | Month 1 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
The Bayley Scales of Infant Development, 4th edition | Month 2 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
The Bayley Scales of Infant Development, 4th edition | Month 3 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
The Bayley Scales of Infant Development, 4th edition | Month 4 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
The Bayley Scales of Infant Development, 4th edition | Month 5 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
The Bayley Scales of Infant Development, 4th edition | Month 6 of infant's life
  The Bayley-4 is a standardized, norm-referenced tool with subtest level scaled scores, domain level composite scores, percentile ranks, and developmental age equivalents. The investigators will utilize the cognitive and motor sections only for this study. The purpose of this outcome measure is to compare developmental trajectories over the first six months of life between the three groups (supervised exercise group, home exercise group, and control group). The highest possible score on a subtest or subdomain is 19, and the lowest possible score is 1. Scores from 8-12 are considered average.
Balke-Ware Submaximal Test | Baseline (late first trimester)
  Used to estimate cardiovascular condition and endurance by measuring maximum oxygen uptake, known as VO2max. Comparison of the participant's heart rate and blood pressure response to exercise between measurements will assess the effect of the intervention on the participant's aerobic capacity. A reduction in heart rate or blood pressure may be consistent with improved aerobic conditioning.
Balke-Ware Submaximal Test | 3 months post-delivery
  Used to estimate cardiovascular condition and endurance by measuring maximum oxygen uptake, known as VO2max. Comparison of the participant's heart rate and blood pressure response to exercise between measurements will assess the effect of the intervention on the participant's aerobic capacity. A reduction in heart rate or blood pressure may be consistent with improved aerobic conditioning.
Balke-Ware Submaximal Test | 6 months post-delivery
  Used to estimate cardiovascular condition and endurance by measuring maximum oxygen uptake, known as VO2max. Comparison of the participant's heart rate and blood pressure response to exercise between measurements will assess the effect of the intervention on the participant's aerobic capacity. A reduction in heart rate or blood pressure may be consistent with improved aerobic conditioning.

SECONDARY OUTCOMES:
Short From-12 Generic Quality of Life | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  A self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The United States population average PCS-12 and MCS-12 are both 50 points.
Multidimensional Fatigue Inventory | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  A 20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Higher total scores correspond with more acute levels of fatigue.
Pittsburgh Sleep Quality Index | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Possible range of scores is 0 to 21, with higher scores indicating worse sleep quality.
Center for Epidemiologic Studies Depression Scale | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  A 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
Edinburgh Postnatal Depression Scale | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  Evaluates whether a woman has symptoms of depression and anxiety during pregnancy and in the year following the birth of a child. Possible range of scores is 0 to 30. Mothers scoring above 12 are likely to be suffering from depression.
Pregnancy Physical Activity Questionnaire | Baseline (late first trimester), late second trimester (25-26 weeks), late third trimester (37-38 weeks), and monthly through 6-months post-natal
  Self-administered semiquantitative questionnaire for assessing typical physical activity, occupational activity, and home activity completed. From the questionnaire, the number of hours spent in each activity is multiplied by the activity intensity to arrive at a measure of average daily energy expenditure (MET-hours per day) attributable to each activity.
Height | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6 of infant's life
  Infant height in centimeters
Weight | Month 1, Month 2, Month 3, Month 4, Month 5, Month 6 of infant's life
  Infant weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Erin Wentz, PT, PhD, Principal Investigator — State University of New York - Upstate Medical University; Carol Sames, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
Because this information is a feasibility study, the investigators will continue to use this study to apply for future grants and it is not possible to determine when this will be complete.

REFERENCES:
- [Background] Evenson KR, Wen F. Prevalence and correlates of objectively measured physical activity and sedentary behavior among US pregnant women. Prev Med. 2011 Jul-Aug;53(1-2):39-43. doi: 10.1016/j.ypmed.2011.04.014. Epub 2011 May 4. PMID 21575654
- [Background] Jukic A MZ, Evenson KR, Herring AH, Wilcox AJ, Hartmann KE, Daniels JL. Correlates of physical activity at two time points during pregnancy. J Phys Act Health. 2012 Mar;9(3):325-35. doi: 10.1123/jpah.9.3.325. PMID 22454434
- [Background] Santo EC, Forbes PW, Oken E, Belfort MB. Determinants of physical activity frequency and provider advice during pregnancy. BMC Pregnancy Childbirth. 2017 Sep 5;17(1):286. doi: 10.1186/s12884-017-1460-z. PMID 28870169
- [Background] Nascimento SL, Surita FG, Cecatti JG. Physical exercise during pregnancy: a systematic review. Curr Opin Obstet Gynecol. 2012 Dec;24(6):387-94. doi: 10.1097/GCO.0b013e328359f131. PMID 23014142
- [Background] Kramer MS. Aerobic exercise for women during pregnancy. Cochrane Database Syst Rev. 2002;(2):CD000180. doi: 10.1002/14651858.CD000180. PMID 12076383
- [Background] Ramirez-Velez R, Aguilar de Plata AC, Escudero MM, Echeverry I, Ortega JG, Salazar B, Rey JJ, Hormiga C, Lopez-Jaramillo P. Influence of regular aerobic exercise on endothelium-dependent vasodilation and cardiorespiratory fitness in pregnant women. J Obstet Gynaecol Res. 2011 Nov;37(11):1601-8. doi: 10.1111/j.1447-0756.2011.01582.x. Epub 2011 Jul 6. PMID 21733037
- [Background] Hegaard HK, Pedersen BK, Nielsen BB, Damm P. Leisure time physical activity during pregnancy and impact on gestational diabetes mellitus, pre-eclampsia, preterm delivery and birth weight: a review. Acta Obstet Gynecol Scand. 2007;86(11):1290-6. doi: 10.1080/00016340701647341. Epub 2007 Sep 7. PMID 17851805
- [Background] Muktabhant B, Lawrie TA, Lumbiganon P, Laopaiboon M. Diet or exercise, or both, for preventing excessive weight gain in pregnancy. Cochrane Database Syst Rev. 2015 Jun 15;2015(6):CD007145. doi: 10.1002/14651858.CD007145.pub3. PMID 26068707
- [Background] Robledo-Colonia AF, Sandoval-Restrepo N, Mosquera-Valderrama YF, Escobar-Hurtado C, Ramirez-Velez R. Aerobic exercise training during pregnancy reduces depressive symptoms in nulliparous women: a randomised trial. J Physiother. 2012;58(1):9-15. doi: 10.1016/S1836-9553(12)70067-X. PMID 22341377
- [Background] Baker JH, Rothenberger SD, Kline CE, Okun ML. Exercise during early pregnancy is associated with greater sleep continuity. Behav Sleep Med. 2018 Sep-Oct;16(5):482-493. doi: 10.1080/15402002.2016.1228649. Epub 2016 Oct 14. PMID 27739877
- [Background] Krzepota J, Sadowska D, Biernat E. Relationships between Physical Activity and Quality of Life in Pregnant Women in the Second and Third Trimester. Int J Environ Res Public Health. 2018 Dec 5;15(12):2745. doi: 10.3390/ijerph15122745. PMID 30563083
- [Background] Kolomanska-Bogucka D, Mazur-Bialy AI. Physical Activity and the Occurrence of Postnatal Depression-A Systematic Review. Medicina (Kaunas). 2019 Sep 2;55(9):560. doi: 10.3390/medicina55090560. PMID 31480778
- [Background] Wiebe HW, Boule NG, Chari R, Davenport MH. The effect of supervised prenatal exercise on fetal growth: a meta-analysis. Obstet Gynecol. 2015 May;125(5):1185-1194. doi: 10.1097/AOG.0000000000000801. PMID 25932847
- [Background] McMillan AG, May LE, Gaines GG, Isler C, Kuehn D. Effects of Aerobic Exercise during Pregnancy on 1-Month Infant Neuromotor Skills. Med Sci Sports Exerc. 2019 Aug;51(8):1671-1676. doi: 10.1249/MSS.0000000000001958. PMID 30817721
- [Background] Davenport MH, McCurdy AP, Mottola MF, Skow RJ, Meah VL, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Riske L, Sobierajski F, James M, Nagpal T, Marchand AA, Nuspl M, Slater LG, Barakat R, Adamo KB, Davies GA, Ruchat SM. Impact of prenatal exercise on both prenatal and postnatal anxiety and depressive symptoms: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1376-1385. doi: 10.1136/bjsports-2018-099697. PMID 30337464
- [Background] Davenport MH, Ruchat SM, Poitras VJ, Jaramillo Garcia A, Gray CE, Barrowman N, Skow RJ, Meah VL, Riske L, Sobierajski F, James M, Kathol AJ, Nuspl M, Marchand AA, Nagpal TS, Slater LG, Weeks A, Adamo KB, Davies GA, Barakat R, Mottola MF. Prenatal exercise for the prevention of gestational diabetes mellitus and hypertensive disorders of pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1367-1375. doi: 10.1136/bjsports-2018-099355. PMID 30337463
- [Background] Davenport MH, Meah VL, Ruchat SM, Davies GA, Skow RJ, Barrowman N, Adamo KB, Poitras VJ, Gray CE, Jaramillo Garcia A, Sobierajski F, Riske L, James M, Kathol AJ, Nuspl M, Marchand AA, Nagpal TS, Slater LG, Weeks A, Barakat R, Mottola MF. Impact of prenatal exercise on neonatal and childhood outcomes: a systematic review and meta-analysis. Br J Sports Med. 2018 Nov;52(21):1386-1396. doi: 10.1136/bjsports-2018-099836. PMID 30337465
- [Background] Campolong K, Jenkins S, Clark MM, Borowski K, Nelson N, Moore KM, Bobo WV. The association of exercise during pregnancy with trimester-specific and postpartum quality of life and depressive symptoms in a cohort of healthy pregnant women. Arch Womens Ment Health. 2018 Apr;21(2):215-224. doi: 10.1007/s00737-017-0783-0. Epub 2017 Oct 24. PMID 29067551
- [Background] Bediako PT, BeLue R, Hillemeier MM. A Comparison of Birth Outcomes Among Black, Hispanic, and Black Hispanic Women. J Racial Ethn Health Disparities. 2015 Dec;2(4):573-82. doi: 10.1007/s40615-015-0110-2. Epub 2015 Apr 23. PMID 26561541
- [Background] Mutambudzi M, Meyer JD, Reisine S, Warren N. A review of recent literature on materialist and psychosocial models for racial and ethnic disparities in birth outcomes in the US, 2000-2014. Ethn Health. 2017 Jun;22(3):311-332. doi: 10.1080/13557858.2016.1247150. Epub 2016 Nov 16. PMID 27852109
- [Background] Christian LM. At the forefront of psychoneuroimmunology in pregnancy: Implications for racial disparities in birth outcomes PART 1: Behavioral risks factors. Neurosci Biobehav Rev. 2020 Oct;117:319-326. doi: 10.1016/j.neubiorev.2019.04.009. Epub 2019 Apr 18. PMID 31005626
- [Background] Gaston A, Cramp A. Exercise during pregnancy: a review of patterns and determinants. J Sci Med Sport. 2011 Jul;14(4):299-305. doi: 10.1016/j.jsams.2011.02.006. Epub 2011 Mar 21. PMID 21420359
- [Background] Di Mascio D, Magro-Malosso ER, Saccone G, Marhefka GD, Berghella V. Exercise during pregnancy in normal-weight women and risk of preterm birth: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Nov;215(5):561-571. doi: 10.1016/j.ajog.2016.06.014. Epub 2016 Jun 16. PMID 27319364
- [Background] Barakat R, Pelaez M, Cordero Y, Perales M, Lopez C, Coteron J, Mottola MF. Exercise during pregnancy protects against hypertension and macrosomia: randomized clinical trial. Am J Obstet Gynecol. 2016 May;214(5):649.e1-8. doi: 10.1016/j.ajog.2015.11.039. Epub 2015 Dec 15. PMID 26704894
- [Background] da Silva SG, Ricardo LI, Evenson KR, Hallal PC. Leisure-Time Physical Activity in Pregnancy and Maternal-Child Health: A Systematic Review and Meta-Analysis of Randomized Controlled Trials and Cohort Studies. Sports Med. 2017 Feb;47(2):295-317. doi: 10.1007/s40279-016-0565-2. PMID 27282925
- [Background] Tobias DK, Zhang C, van Dam RM, Bowers K, Hu FB. Physical activity before and during pregnancy and risk of gestational diabetes mellitus: a meta-analysis. Diabetes Care. 2011 Jan;34(1):223-9. doi: 10.2337/dc10-1368. Epub 2010 Sep 27. PMID 20876206
- [Background] Aune D, Saugstad OD, Henriksen T, Tonstad S. Maternal body mass index and the risk of fetal death, stillbirth, and infant death: a systematic review and meta-analysis. JAMA. 2014 Apr 16;311(15):1536-46. doi: 10.1001/jama.2014.2269. PMID 24737366
- [Background] Streuling I, Beyerlein A, Rosenfeld E, Hofmann H, Schulz T, von Kries R. Physical activity and gestational weight gain: a meta-analysis of intervention trials. BJOG. 2011 Feb;118(3):278-84. doi: 10.1111/j.1471-0528.2010.02801.x. Epub 2010 Dec 7. PMID 21134106
- [Background] Vargas-Terrones M, Barakat R, Santacruz B, Fernandez-Buhigas I, Mottola MF. Physical exercise programme during pregnancy decreases perinatal depression risk: a randomised controlled trial. Br J Sports Med. 2019 Mar;53(6):348-353. doi: 10.1136/bjsports-2017-098926. Epub 2018 Jun 13. PMID 29899050
- [Background] Goodwin A, Astbury J, McMeeken J. Body image and psychological well-being in pregnancy. A comparison of exercisers and non-exercisers. Aust N Z J Obstet Gynaecol. 2000 Nov;40(4):442-7. doi: 10.1111/j.1479-828x.2000.tb01178.x. PMID 11194433
- [Background] Chan CWH, Au Yeung E, Law BMH. Effectiveness of Physical Activity Interventions on Pregnancy-Related Outcomes among Pregnant Women: A Systematic Review. Int J Environ Res Public Health. 2019 May 23;16(10):1840. doi: 10.3390/ijerph16101840. PMID 31126153
- [Background] Haakstad LA, Bo K. Exercise in pregnant women and birth weight: a randomized controlled trial. BMC Pregnancy Childbirth. 2011 Sep 30;11:66. doi: 10.1186/1471-2393-11-66. PMID 21961534
- [Background] Vega SR, Kleinert J, Sulprizio M, Hollmann W, Bloch W, Struder HK. Responses of serum neurotrophic factors to exercise in pregnant and postpartum women. Psychoneuroendocrinology. 2011 Feb;36(2):220-7. doi: 10.1016/j.psyneuen.2010.07.012. Epub 2010 Aug 6. PMID 20692101
- [Background] Labonte-Lemoyne E, Curnier D, Ellemberg D. Exercise during pregnancy enhances cerebral maturation in the newborn: A randomized controlled trial. J Clin Exp Neuropsychol. 2017 May;39(4):347-354. doi: 10.1080/13803395.2016.1227427. Epub 2016 Sep 13. PMID 27622854
- [Background] Hopkins SA, Cutfield WS. Exercise in pregnancy: weighing up the long-term impact on the next generation. Exerc Sport Sci Rev. 2011 Jul;39(3):120-7. doi: 10.1097/JES.0b013e31821a5527. PMID 21519301
- [Background] Lewis BA, Schuver K, Dunsiger S, Samson L, Frayeh AL, Terrell CA, Ciccolo JT, Avery MD. Rationale, design, and baseline data for the Healthy Mom II Trial: A randomized trial examining the efficacy of exercise and wellness interventions for the prevention of postpartum depression. Contemp Clin Trials. 2018 Jul;70:15-23. doi: 10.1016/j.cct.2018.05.002. Epub 2018 May 7. PMID 29747048
- [Background] Shakeel N, Richardsen KR, Martinsen EW, Eberhard-Gran M, Slinning K, Jenum AK. Physical activity in pregnancy and postpartum depressive symptoms in a multiethnic cohort. J Affect Disord. 2018 Aug 15;236:93-100. doi: 10.1016/j.jad.2018.04.081. Epub 2018 Apr 23. PMID 29723768
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Sexton MB, Flynn HA, Lancaster C, Marcus SM, McDonough SC, Volling BL, Lopez JF, Kaciroti N, Vazquez DM. Predictors of recovery from prenatal depressive symptoms from pregnancy through postpartum. J Womens Health (Larchmt). 2012 Jan;21(1):43-9. doi: 10.1089/jwh.2010.2266. Epub 2011 Nov 7. PMID 22060255
- [Background] Coll CV, Domingues MR, Goncalves H, Bertoldi AD. Perceived barriers to leisure-time physical activity during pregnancy: A literature review of quantitative and qualitative evidence. J Sci Med Sport. 2017 Jan;20(1):17-25. doi: 10.1016/j.jsams.2016.06.007. Epub 2016 Jun 23. PMID 27372276
- [Background] Evenson KR, Moos MK, Carrier K, Siega-Riz AM. Perceived barriers to physical activity among pregnant women. Matern Child Health J. 2009 May;13(3):364-75. doi: 10.1007/s10995-008-0359-8. Epub 2008 May 14. PMID 18478322
- [Background] ACOG Committee Opinion No. 650: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstet Gynecol. 2015 Dec;126(6):e135-e142. doi: 10.1097/AOG.0000000000001214. PMID 26595585
- [Background] Pollock ML, Foster C, Schmidt D, Hellman C, Linnerud AC, Ward A. Comparative analysis of physiologic responses to three different maximal graded exercise test protocols in healthy women. Am Heart J. 1982 Mar;103(3):363-73. doi: 10.1016/0002-8703(82)90275-7. PMID 7064770
- [Background] Emmanuel E, St John W, Sun J. Relationship between social support and quality of life in childbearing women during the perinatal period. J Obstet Gynecol Neonatal Nurs. 2012 Nov-Dec;41(6):E62-70. doi: 10.1111/j.1552-6909.2012.01400.x. Epub 2012 Aug 3. PMID 22861382
- [Background] Fisher J, Wynter K, Hammarberg K, McBain J, Gibson F, Boivin J, McMahon C. Age, mode of conception, health service use and pregnancy health: a prospective cohort study of Australian women. BMC Pregnancy Childbirth. 2013 Apr 8;13:88. doi: 10.1186/1471-2393-13-88. PMID 23565589
- [Background] De Pascalis L, Agostini F, Monti F, Paterlini M, Fagandini P, La Sala GB. A comparison of quality of life following spontaneous conception and assisted reproduction. Int J Gynaecol Obstet. 2012 Sep;118(3):216-9. doi: 10.1016/j.ijgo.2012.04.020. Epub 2012 Jun 22. PMID 22727413
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Beeghly M, Olson KL, Weinberg MK, Pierre SC, Downey N, Tronick EZ. Prevalence, stability, and socio-demographic correlates of depressive symptoms in Black mothers during the first 18 months postpartum. Matern Child Health J. 2003 Sep;7(3):157-68. doi: 10.1023/a:1025132320321. PMID 14509411
- [Background] Boyd RC, Le HN, Somberg R. Review of screening instruments for postpartum depression. Arch Womens Ment Health. 2005 Sep;8(3):141-53. doi: 10.1007/s00737-005-0096-6. Epub 2005 Sep 5. PMID 16133785
- [Background] Campbell SB, Cohn JF. Prevalence and correlates of postpartum depression in first-time mothers. J Abnorm Psychol. 1991 Nov;100(4):594-9. doi: 10.1037//0021-843x.100.4.594. PMID 1757673
- [Background] Davies GA, Wolfe LA, Mottola MF, MacKinnon C; Society of Obstetricians and gynecologists of Canada, SOGC Clinical Practice Obstetrics Committee. Joint SOGC/CSEP clinical practice guideline: exercise in pregnancy and the postpartum period. Can J Appl Physiol. 2003 Jun;28(3):330-41. PMID 12955862
- [Background] Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004 Oct;36(10):1750-60. doi: 10.1249/01.mss.0000142303.49306.0d. PMID 15595297
- [Background] Bamfo JE, Kametas NA, Nicolaides KH, Chambers JB. Maternal left ventricular diastolic and systolic long-axis function during normal pregnancy. Eur J Echocardiogr. 2007 Oct;8(5):360-8. doi: 10.1016/j.euje.2006.12.004. Epub 2007 Feb 23. PMID 17321800
- [Background] Naqvi TZ, Elkayam U. Serial echocardiographic assessment of the human heart in normal pregnancy. Circ Cardiovasc Imaging. 2012 May 1;5(3):283-5. doi: 10.1161/CIRCIMAGING.112.974808. No abstract available. PMID 22592007
- [Background] van Delft K, Schwertner-Tiepelmann N, Thakar R, Sultan AH. Recruitment of pregnant women in research. J Obstet Gynaecol. 2013 Jul;33(5):442-6. doi: 10.3109/01443615.2013.767787. PMID 23815192
- [Background] Carpenter RE, Emery SJ, Rassi D, Uzun O, Lewis MJ. Recruitment of pregnant women to an exercise-intervention study. J Obstet Gynaecol. 2016;36(2):200-7. doi: 10.3109/01443615.2015.1049988. Epub 2015 Oct 14. PMID 26467417
- See also: Census bureau statistics for Syracuse — https://www.census.gov/quickfacts/fact/table/syracusecitynewyork/IPE120218

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT05394883/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT05394883/ICF_001.pdf